CLINICAL TRIAL: NCT01588873
Title: The Effects of Contraceptive Pill and Hormonal Vaginal Ring on Hormonal, Inflammatory and Metabolic Parameters in Women of Reproductive Age With Polycystic Ovary Syndrome (PCOS).
Brief Title: Contraceptive Pill and Hormonal Vaginal Ring in Women With Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 106/2011
Record Dates: First submitted 2012-03-28; First posted 2012-05-01 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Adverse Effect of Oral Contraceptives, Sequela
Keywords: Oral contraceptive pill; Hormonal contraceptive ring; Polycystic ovary syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — ethinyl estradiol-desogestrel combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral contraceptive pill (Active Comparator)
  Interventions: Drug: oc:E-E-desogestrel/vaginal ring:E-E -ethonogestrel
- Contraceptive ring (Active Comparator)
  Interventions: Drug: oc:E-E-desogestrel/vaginal ring:E-E -ethonogestrel

INTERVENTIONS:
Drug: oc:E-E-desogestrel/vaginal ring:E-E -ethonogestrel — The OC or vaginal ring will be used in 9 weeks periods followed by one week's break each.
  After a wash-out period of at least 2 months of any previous hormonal contraceptives all examinations will be performed at the 1st to 5th day of the menstruation cycle at baseline and then at the 9th, 29th and 59th week and the last 1 month after stopping contraception.
  Blood samples will be collected between 07 and 10 AM after an overnight fast and during the follicular phase or at any time in cases of amenorrhea. After centrifugation serum is filled in eight tubes with at least 2 ml of serum in each, and immediately frozen at -70ºC as well as one tube of plasma. Every tube will be marked appropriately. Fasting plasma glucose and HbA1c will be analysed at once at every appointment.
  Other Names: Mercilon, Nuva-Ring

SUMMARY:
The main aims of this study are:

* to investigate and compare the effects of long lasting use (59 weeks) of vaginal and oral contraceptives on androgen secretion, insulin and glucose metabolism, lipid profile, and serum levels of SHBG and hs-CRP in women with PCOS.
* to compare the metabolic effects of oral and vaginal combined contraceptives and to find out whether oral or transvaginal contraceptive can be recommended to a particular group of women, for example in women with increased metabolic risks.
* to clarify whether the unfavourable effects of combined contraceptives diminish with time (after use of one year).

DETAILED DESCRIPTION:
The study population consists of women of reproductive age with PCOS, no wish of pregnancy and no other contraindications to hormonal contraceptives.

The volunteer subjects will be recruited from hospital's patient files with PCOS (IC diagnosis E.28.2).

Methods Sample size Our previous study comparing the metabolic effects of the same preparations (Mercilon and Nuvaring) in young healthy women shown an significant decrease of 1.65 (SD 1.68)in the Matsuda index at 9 weeks of treatment with oral contraceptive pill. Power analysis indicated that 14 women would be needed in both groups to reveal a similar significant decrease in the serum level of Matsuda index. To allow for drop-outs (estimated to be as high as 20-30%), the planned sample size will be 21 in each group.

Medication Forty women will be randomised either to the pill (n=21) or ring (n=21) group. The OC or contraceptive ring will be used in nine weeks periods. Every period will be followed by a break of one week.

In the pill group the subjects start the pill during the first days of the follicular phase of the cycle after the baseline examinations and continue nonstop for nine weeks, i.e. until the third package has ran out. This is followed by one weeks' break. The ring is replaced every three weeks and the treatment is continued nine weeks after which one week break follows. In both groups the cycle will be repeated six times resulting in 59 weeks of treatment.

The used preparations are: Vaginal ring, depotproduct: ethinylestradiol 2.7 mg (0,015 mg/day) and etonogestrel 11.7 mg (0,120 mg/day)and the contraceptive pill, ethinylestradiol tabl 20 µg, desogestrel 150 µg.

Ultrasonography An ultrasonography of the ovaries will be performed at baseline to support the diagnosis of PCOS and exclude any androgen releasing tumors.

Blood samples Blood samples for hormonal and metabolic assessments will be taken at every appointment.

Oral glucose tolerance test (OGTT) The glucose metabolism and tolerance are measured with an oral glucose tolerance test, where the subjects take a dose of 75 grams of glucose mixed in 300ml of water after ten hours fasting. The blood samples are taken before the test and 30, 60 and 120 minutes after the glucose intake.

The schedule A wash-out period of at least 2 months after the use of any previous hormonal contraceptives will be required. At baseline all examinations are performed at the 1st to 5th day of the menstruation cycle before beginning contraception.

The second appointment will occur during the 9th pill/ring week, the third at the 29th week, the fourth at the 59th week and the last appointment one month after stopping contraception. Blood samples are taken and blood pressure is measured at every appointment, OGTT will be performed at every appointment except at the 29th week.

Serum analyses All blood samples will be collected in the morning between 07 and 10 after an overnight fast and during the follicular phase (cycle days 1-4) or at any time in cases of amenorrhea. All screening analyses will be analysed at the local hospital.

Seven test-tubes whole blood are collected from each patient. Six tubes are centrifuged within 30 minutes, and serum is filled in eight (8) tubes with at least 2 ml of serum in each, and immediately frozen at -70 º C. In addition, the plasma from one tube will frozen at -70 º C in at least 2 tubes with at least 2ml plasma in each. Every tube is marked by randomisation number, initials, date of birth and time.

Fasting plasma glucose and HbA1c will be analysed at once at every appointment at the local hospital.

Planned analyses Hormonal, metabolic and inflammatory parameters. Ethical questions and possible harmful effects Participating in the research is completely voluntary. When taking the blood samples, the risks are practically restricted to the problems caused by the stitch of the needle.

The possible adverse effects of the used contraceptives are observed at every appointment. Problems are reported to FIMEA (Finnish Medical Association) and to the local ethical committee, if necessary.

A continuous dosing is used in this study, which is not routine treatment. Uninterrupted dosing of contraceptive pills has been used in several studies and no differences in the contraceptive effect compared to routine dosing have been reported. Instead, the menstruation comes less frequently which is user-friendly. Continuous dosing may cause slightly more swelling and extra leakage.

After the study the treatment of the subjects continues following standard practice.

All information required will be kept locked in cupboards, and disposed ten years after the study has ended. Information on computer requires username and password.

Analysing the results and their significance Blood samples are analyzed in Oulu University Hospital laboratory of Clinical Chemistry, which fulfills international quality criteria. The results are analyzed using SPSS-program. During the research Oulu University statistics-professional will be consulted for help in the statistical analyses.

Significance of the study:

This study will allow to clarify whether oral or transvaginal contraceptive can be recommended to a particular group of women, for example in women with increased metabolic risks. It will also clarify whether the unfavourable effects of combined contraceptives decrease after long term use.

Concealment and disposing the register The information and study data will be kept on computer requiring a username and password. All written information will be kept in a room in locked cupboards. The register will be disposed following ethical committee's instructions no later than the end of 2027.

Schedule The study will begin in spring 2012 and is estimated to continue until December 2018.

Funding The study will be funded by the Sigrid Juselius organization and from the Kevo-fund of Department of Obstetrics and Gynaecology of Oulu University Hospital.

Changes in the plan Every possible changes in the study design will be reported to the local Ethical Committee.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 18 to 40 years
* diagnosed PCOS (Rotterdam criteria)
* healthy, no medications
* no use of hormonal contraceptives or wash-out period of at least two months
* no contraindications to hormonal contraception

Exclusion Criteria:

* regular smoking
* excessive alcohol use
* pregnancy or breastfeeding
* oversensitivity to active ingredients
* migraine with focal aura
* severe or multiple risk factors to thrombosis
* diagnosed or suspected cancer
* diagnosed or suspected estrogen-dependent tumor
* acute or chronic hepatocellular disease -related abnormal liver function
* hepatic adenomas or carcinomas
* undiagnosed abnormal vaginal bleeding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2012-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in Matsuda index during the oral contraceptive pill (E-E-desogestrel)/vaginal ring (E-E -ethonogestrel) | Change from baseline in Matsuda index at 59 weeks of treament
  Calculation of the Matsuda index according to the following equation: [10000 / √((fasting glucose x fasting insulin)x (Gmeanogtt x Imeanogtt))]

SECONDARY OUTCOMES:
Change in high sensitive C-reactive protein (mg/l) during the oral contraceptive pill (E-E-desogestrel)/vaginal ring (E-E -ethonogestrel) | Change from baseline in serum CRP concentrations at 59 weeks of treament
Change in Free Androgen Index during the oral contraceptive pill (E-E-desogestrel)/vaginal ring (E-E -ethonogestrel) | Change from baseline in Free Androgen Index at 59 weeks of treament
  Calculation by using the equation 100×T (nmol/l)/SHBG (nmol/l).

CONTACTS AND LOCATIONS:
Overall Officials: Laure C Morin-Papunen, Principal Investigator — University of Oulu
Locations (1):
- Department of Obstetrics and Gynaecology, University Hospital of Oulu, Oulu, Finland

REFERENCES:
- [Background] Acien P, Mauri M, Gutierrez M. Clinical and hormonal effects of the combination gonadotrophin-releasing hormone agonist plus oral contraceptive pills containing ethinyl-oestradiol (EE) and cyproterone acetate (CPA) versus the EE-CPA pill alone on polycystic ovarian disease-related hyperandrogenisms. Hum Reprod. 1997 Mar;12(3):423-9. doi: 10.1093/humrep/12.3.423. PMID 9130733
- [Background] Allen HF, Mazzoni C, Heptulla RA, Murray MA, Miller N, Koenigs L, Reiter EO. Randomized controlled trial evaluating response to metformin versus standard therapy in the treatment of adolescents with polycystic ovary syndrome. J Pediatr Endocrinol Metab. 2005 Aug;18(8):761-8. doi: 10.1515/jpem.2005.18.8.761. PMID 16200842
- [Background] Armstrong VL, Wiggam MI, Ennis CN, Sheridan B, Traub AI, Atkinson AB, Bell PM. Insulin action and insulin secretion in polycystic ovary syndrome treated with ethinyl oestradiol/cyproterone acetate. QJM. 2001 Jan;94(1):31-7. doi: 10.1093/qjmed/94.1.31. PMID 11161134
- [Background] Ball MJ, Ashwell E, Jackson M, Gillmer MD. Comparison of two triphasic contraceptives with different progestogens: effects on metabolism and coagulation proteins. Contraception. 1990 Apr;41(4):363-76. doi: 10.1016/0010-7824(90)90036-u. PMID 2335101
- [Background] Bilgir O, Kebapcilar L, Taner C, Bilgir F, Kebapcilar A, Bozkaya G, Yildiz Y, Yuksel A, Sari I. The effect of ethinylestradiol (EE)/cyproterone acetate (CA) and EE/CA plus metformin treatment on adhesion molecules in cases with polycystic ovary syndrome (PCOS). Intern Med. 2009;48(14):1193-9. doi: 10.2169/internalmedicine.48.2177. Epub 2009 Jul 15. PMID 19602786
- [Background] Cagnacci A, Paoletti AM, Renzi A, Orru M, Pilloni M, Melis GB, Volpe A. Glucose metabolism and insulin resistance in women with polycystic ovary syndrome during therapy with oral contraceptives containing cyproterone acetate or desogestrel. J Clin Endocrinol Metab. 2003 Aug;88(8):3621-5. doi: 10.1210/jc.2003-030328. PMID 12915645
- [Background] Carranza-Lira S, Magana-Padilla NR. [Ultrasonographic and lipid changes in polycystic ovary syndrome according to the type of treatment ]. Ginecol Obstet Mex. 2002 Jun;70:285-8. Spanish. PMID 12148471
- [Background] Charitidou C, Farmakiotis D, Zournatzi V, Pidonia I, Pegiou T, Karamanis N, Hatzistilianou M, Katsikis I, Panidis D. The administration of estrogens, combined with anti-androgens, has beneficial effects on the hormonal features and asymmetric dimethyl-arginine levels, in women with the polycystic ovary syndrome. Atherosclerosis. 2008 Feb;196(2):958-65. doi: 10.1016/j.atherosclerosis.2007.03.002. Epub 2007 Apr 6. PMID 17418849
- [Background] Chasan-Taber L, Willett WC, Stampfer MJ, Hunter DJ, Colditz GA, Spiegelman D, Manson JE. A prospective study of oral contraceptives and NIDDM among U.S. women. Diabetes Care. 1997 Mar;20(3):330-5. doi: 10.2337/diacare.20.3.330. PMID 9051382
- [Background] Chen MJ, Yang WS, Chen HF, Kuo JJ, Ho HN, Yang YS, Chen SU. Increased follistatin levels after oral contraceptive treatment in obese and non-obese women with polycystic ovary syndrome. Hum Reprod. 2010 Mar;25(3):779-85. doi: 10.1093/humrep/dep459. Epub 2010 Jan 20. PMID 20093255
- [Background] Cibula D, Sindelka G, Hill M, Fanta M, Skrha J, Zivny J. Insulin sensitivity in non-obese women with polycystic ovary syndrome during treatment with oral contraceptives containing low-androgenic progestin. Hum Reprod. 2002 Jan;17(1):76-82. doi: 10.1093/humrep/17.1.76. PMID 11756365
- [Background] Cibula D, Fanta M, Vrbikova J, Stanicka S, Dvorakova K, Hill M, Skrha J, Zivny J, Skrenkova J. The effect of combination therapy with metformin and combined oral contraceptives (COC) versus COC alone on insulin sensitivity, hyperandrogenaemia, SHBG and lipids in PCOS patients. Hum Reprod. 2005 Jan;20(1):180-4. doi: 10.1093/humrep/deh588. Epub 2004 Dec 2. PMID 15576394
- [Background] Costello MF, Shrestha B, Eden J, Johnson NP, Sjoblom P. Metformin versus oral contraceptive pill in polycystic ovary syndrome: a Cochrane review. Hum Reprod. 2007 May;22(5):1200-9. doi: 10.1093/humrep/dem005. Epub 2007 Jan 29. PMID 17261574
- [Background] Creatsas G, Koliopoulos C, Mastorakos G. Combined oral contraceptive treatment of adolescent girls with polycystic ovary syndrome. Lipid profile. Ann N Y Acad Sci. 2000;900:245-52. doi: 10.1111/j.1749-6632.2000.tb06236.x. PMID 10818412
- [Background] Duleba AJ, Banaszewska B, Spaczynski RZ, Pawelczyk L. Simvastatin improves biochemical parameters in women with polycystic ovary syndrome: results of a prospective, randomized trial. Fertil Steril. 2006 Apr;85(4):996-1001. doi: 10.1016/j.fertnstert.2005.09.030. Epub 2006 Mar 9. PMID 16580386
- [Background] Dunaif A, Segal KR, Futterweit W, Dobrjansky A. Profound peripheral insulin resistance, independent of obesity, in polycystic ovary syndrome. Diabetes. 1989 Sep;38(9):1165-74. doi: 10.2337/diab.38.9.1165. PMID 2670645
- [Background] Ehrmann DA. Polycystic ovary syndrome. N Engl J Med. 2005 Mar 24;352(12):1223-36. doi: 10.1056/NEJMra041536. No abstract available. PMID 15788499